CLINICAL TRIAL: NCT05577507
Title: Efficacy and Safety of Cholestyramine in the Management of Hyperphosphatemia in Adult Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Essam Aly, Demonstrator at clinical pharmacy department , Sinai university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC#102
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Hemodialysis Complication; Hyperphosphatemia
Keywords: chronic kidney disease; hyperphosphatemia in chronic adult hemodialysis patients; bile acid sequestrants: cholestyramine; serum calcium level, serum phosphate level
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — Cholestyramine Resin; Calcium Carbonate; Tablets

STUDY DESIGN:
Intervention Model Description: A total of 80 patients will be recruited and divided into 2 groups: -
  Group 1: (cholestyramine 12 gram), 40 patients will take a dose of cholestyramine 4-gram sachet three times daily with standard therapy(Calcimate).
  Group 2: Control group, 40 patients will take only the standard therapy (Calcimate).
  Time of the trial will be two months (8 weeks trial period)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Active Comparator): Group 1:
  (cholestyramine 12 gram), 40 patients will take a dose of cholestyramine 4-gram sachets three times daily within meals with (Calcimate).
  Dosage: one sachet on 150 ml water three times daily duration : 8 weeks
  Interventions: Drug: Cholestyramine Resin 4000 MG [Questran]; Drug: Calcium Carbonate 500 MG Oral Tablet
- Control group (Placebo Comparator): Group 2: Control group, 40 patients will take only (Calcimate).
  Interventions: Drug: Calcium Carbonate 500 MG Oral Tablet

INTERVENTIONS:
Drug: Cholestyramine Resin 4000 MG [Questran] — cholestyramine 4 gram sachets (questran) will be administered orally three times daily for 8 weeks period trial
  Arms: Test group
Drug: Calcium Carbonate 500 MG Oral Tablet — control group will administer standard therapy calcimate 500 mg three times daily within meals

SUMMARY:
After the end of trial, we will examine if cholestyramine has a significant efficacy on reducing serum phosphate level in adult hemodialysis patients.

Time of the trial will be two months (8 weeks trial period)

Baseline characteristics: The following data will be collected from all patients at baseline

1. Age, sex, weight, duration of ESRD and hemodialysis comorbidities.
2. Dialysis duration, serum phosphate level, serum calcium level, iPTH, BUN, Cr (mg/d L), Albumin (mg/d L), Hb (g m%), renal function test, liver function test, blood glucose level, TG, total cholesterol level, LDL-C, HDL.C.

After the end of trial, we will examine if cholestyramine has a significant efficacy on reducing serum phosphate level in adult hemodialysis patients.

DETAILED DESCRIPTION:
Chronic kidney disease-mineral and bone disorder (CKD-MBD) is characterized by progressive loss of renal function as well as dysregulation of mineral and bone metabolism, leading frequently to hyperphosphatemia.

Multiple studies have consistently shown that hyperphosphatemia is associated with cardiovascular events and increased morbidity and mortality in end-stage renal disease (ESRD) patients.

Importantly, use of phosphate binding agents and reduction of serum phosphate concentration are associated with a lower risk of mortality.

The most widely used phosphate binders are calcium-based, although they are frequently associated with hypercalcemia and vascular calcification.

Colestilan is a non-metallic phosphate binder that acts as an anion-exchange resin. Colestilan itself is not absorbed after oral administration, and it is able to bind dietary phosphate within the gastrointestinal tract and thus prevent absorption of the mineral.

A total of 80 patients will be recruited and divided into 2 groups: -

Group 1: 40 patients will take a dose of cholestyramine 4-gram sachet three times daily with standard therapy (Calcimate).

Group 2: 40 patients will take only the standard therapy (Calcimate).

Time of the trial will be two months (8 weeks trial period)

Baseline characteristics: The following data will be collected from all patients at baseline

1. Age, sex, weight, duration of ESRD and hemodialysis comorbidities.
2. Dialysis duration, serum phosphate level, serum calcium level, iPTH, BUN, Cr (mg/d L), Albumin (mg/d L), Hb (g m%), renal function test, liver function test, blood glucose level, TG, total cholesterol level, LDL-C, HDL.C.

After the end of trial, we will examine if cholestyramine has a significant efficacy on reducing serum phosphate level in adult hemodialysis patients.

Parameters will be collected from all patients after 8-week trial period: Serum phosphate, serum calcium, iPTH, LDL, TG and total cholesterol level

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged ≥18 years with CKD stage (4&5)

  * Serum phosphate level ≥ 5.5 mg/dL
  * Serum LDL-C level ≥1.82 mmol/L (70 mg/dL)
  * Hemodialysis frequency 3 times per week or more.
  * Hemodialysis in the last 3 months or longer.

Exclusion Criteria:

* Patients are excluded if they have a history of dysphagia, or swallowing disorder.

  2-patients require warfarin or digoxin treatment. 3- Patients have a history of alcohol or substance abuse 4- Patients receiving calcimimetics. 5- Pregnant patients. 6- Patients have Triglyceride level above 300 (mg/dl)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
serum phosphate level | 8 weeks trial period
  measuring serum phosphate level at baseline and after 8 weeks trial period to evaluate serum phosphate reduction by cholestyramine
serum calcium level | 8 weeks trial period
  measuring serum calcium level at baseline and after 8 weeks trial period to evaluate serum calcium reduction by cholestyramine
iPTH | 8 weeks trial period
  measuring iPTH level at baseline and after 8 weeks trial period to evaluate iPTH reduction by cholestyramine

SECONDARY OUTCOMES:
Lipid Profile ( triglyceride level , LDL ,HDL ,Total cholesterol ) | 8 weeks trial period
  measuring LDL , total cholesterol reduction after using cholestyramine for 8 weeks trial period

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

REFERENCES:
- [Derived] Ghanem AEAEHA, Borolossy RME, Said TWE, Shaheen SMZ. Cholestyramine in hemodialysis: a new approach for hyperphosphatemia management. Korean J Physiol Pharmacol. 2025 Jul 1;29(4):465-473. doi: 10.4196/kjpp.24.269. Epub 2025 Feb 6. PMID 39910709
- See also: Dose of cholestyramine and frequency of administration — https://www.e-enm.org/journal/view.php?doi=10.3803/EnM.2016.31.3.476